CLINICAL TRIAL: NCT01127789
Title: The Use of Transcranial Direct Current Stimulation (tDCS) to Study Implicit Motor Learning on Patients With Brain Injury
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: test device not approved to be used
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 200910005R
Record Dates: First submitted 2010-03-08; First posted 2010-05-21 (Estimated); Last update posted 2012-12-21 (Estimated); Status verified 2012-11

CONDITIONS: Traumatic Brain Injury; Stroke
MeSH Terms: conditions — Brain Injuries, Traumatic; Stroke | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- non-invasive brain stimulation (Experimental)
  Interventions: Device: Transcranial Direct Current Stimulation

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation — Transcranial Direct Current Stimulation
  Other Names: Chanttanooga ionto Dual Channel Stimulator

SUMMARY:
The purpose of this study is to study motor learning and recovery of patients with brain damage caused by traumatic brain injury or stroke with transcranial direct current stimulation (tDCS). It is hypothesized that anodal tDCS on the lesion side and/or cathodal tDCS on the healthy side of motor cortex could improve the recovery of motor function such as learning.

DETAILED DESCRIPTION:
We aim to apply transcranial direct current stimulation (tDCS) to study the recovery process of motor learning on the patients with brain damage caused by traumatic brain injury or stroke. Both anodal and cathodal tDCS will be used to test whether the increase of motor cortical activity by anodal tDCS over lesional side or the decrease of brain activity by cathodal tDCS on healthy side will improve the learning skill (SRTT: serial reaction time task). The result could help to understand the mechanism of motor and cognitive recovery after brain damage, and further rationalize the application of non-invasive brain stimulation such as tDCS for patient rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* TBI or stroke patients
* with partially preserved fine motor function

Exclusion Criteria:

* with metal clips in head or device (e.g. pacemaker)
* with active CNS drugs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-03; Primary Completion 2011-03 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Reaction time (millisecond) | 24 hours post intervention
  Primary outcome measure is the average reaction time of 360 trials from each block -- the task is composed of 8 blocks. After intervention, 3 blocks will be re-tested for 3 times to evaluate the consolidating effect of tDCS on motor learning.

SECONDARY OUTCOMES:
Error rate (percentage) | 24 hours post intervention
  Secondary outcome measure is the error rate of each block which will be re-tested for 3 times after intervention. The aim is to evaluate the motor learning effect during and after tDCS.

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Shiang Chen, MD, PhD, Principal Investigator — Dpt. Physical Medicine and Rehabilitation, NTUH Taipei, Taiwan
Locations (1):
- Dpt. Physical Medicine and Rehabilitation, NTUH, Taipei, Taiwan

REFERENCES:
- [Derived] Elsner B, Kugler J, Pohl M, Mehrholz J. Transcranial direct current stimulation (tDCS) for improving activities of daily living, and physical and cognitive functioning, in people after stroke. Cochrane Database Syst Rev. 2020 Nov 11;11(11):CD009645. doi: 10.1002/14651858.CD009645.pub4. PMID 33175411